CLINICAL TRIAL: NCT06597552
Title: The Effect of Inspiratory Muscle Training on Respiratory Functions, Functional Capacity, Failure and Quailty of Life in Pediatric Cancer Patient
Brief Title: The Effect of Inspiratory Muscle Training on Pediatric Cancer Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Onur Köksal, Assistant Professor, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/001O
Record Dates: First submitted 2024-08-23; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pediatric Cancer; Inspiratory Muscle Training
Keywords: Pediatric Cancer; Inspiratory Muscle Training; Respiratory Function; Muscle Strength
MeSH Terms: conditions — Neoplasms; Respiratory Aspiration | interventions — Sensitivity Training Groups; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistician was blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Other: Control Group
- Training Group (Experimental)
  Interventions: Other: Training Group

INTERVENTIONS:
Other: Training Group — Inspiratory muscle training (IMT) was performed using the Threshold IMT device using the threshold loading method. The IMT was administered to the patients in the training group at 30% of the MIP value, 5 days a week, twice a day, for 15 minutes for 8 weeks. The patients in the training group were called for a check-up once a week and the MIP value was re-evaluated. The training workload for that week was determined by taking 30% of the new measured MIP value.
  During the training, the patients were asked to sit with their upper body (shoulders and upper chest) in a relaxed position, and after the nose was closed with the clip, the mouthpiece of the device was tightly closed with the lips. While in this position, the patient was asked to inhale and exhale 5 times into the device, then remove the device from their mouth and listen for 5 breaths, and continue this cycle for 15 minutes.
  Other Names: Experimental Group
  Arms: Training Group
Other: Control Group — The training intensity of the control group was given at the lowest load (9 cm H2O) for 8 weeks, five days a week, twice a day for 15 minutes. To eliminate the effect of learning, the MIP measure of the control group was measured once a week, but the intensity of the training was not increased during the 8 weeks.
  Arms: Control Group

SUMMARY:
The aim of this study is to examine the effects of inspiratory muscle training on respiratory functions, functional capacity, fatigue and quality of life in pediatric cancer patients who have recently completed treatment. A total of 27 patients were included in the study. The patients were divided into two groups as Training and Control groups. After the initial evaluation of all patients, they were included in an 8-week inspiratory muscle training program. The final evaluation was made at the end of 8 weeks. According to the final evaluations, it was found that there was a statistical increase in favor of the Training group on Maximal Inspiratory Pressure, 6 Minute Walking Test, Quality of Life and Fatigue.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of inspiratory muscle training on respiratory functions, functional capacity, fatigue and quality of life in pediatric cancer patients. A total of 27 patients, 13 in the training group and 14 in the control group, who received and completed cancer treatment at the Memorial Şişli Hospital Pediatric Oncology and Hematology Department and who met the inclusion criteria were included in the study. The age, gender, diagnosis, height and weight of the patients included in the study were recorded. Evaluations were made regarding respiratory functions, respiratory muscle strength, functional capacity, fatigue and quality of life in the patients before and after inspiratory muscle training.

In the study, the initial and post-training values of the FVC, % FVC, FEV1, % FEV1, FEV1/FVC, PEF and % PEF in the respiratory function test of the patients in the training and control groups were compared.

The MIP and MEP values of the patients in the training and control groups were compared with the initial and post-test values of SpO2, heart rate and walking distance calculated after 6MWT. Fatigue values of patients in the education and control groups before and after inspiratory muscle training were compared. Physical, emotional, social and school-related baseline values obtained after the pediatric quality of life test in the education and control groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* Being between 8 and 18 years old
* Having been diagnosed with cancer and having completed treatment
* Having passed at least 30 and at most 120 days after completion of treatment.

Exclusion Criteria:

* Having chronic lung disease,
* Having a history of hospitalization due to infection in the last month,
* Having a history of surgical intervention due to cancer,
* Having insufficient cognitive and cognitive functions,
* Having an orthopedic problem affecting mobility or a history of musculoskeletal surgical intervention,
* Having cancer relapse during the 8-week training program,
* Having received additional chemotherapy for any reason despite having completed treatment,

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Measurement of Pulmonary Function | 8 weeks
  A spirometry device was used to evaluate lung functions and measurements were made according to ATS/ERS criteria. Before the test, the weight (kg), height (cm), age and gender values of the patients were recorded on the spirometry device. All measurements were made in a sitting position with the feet in full contact with the ground. A nose clip was used. At the beginning of the test, inspiration and expiration were requested within the limits of tidal volume. Then, the deepest possible inspiration was followed by rapid expiration. Care was taken to ensure that the expiration period continued uninterrupted for 6 seconds. The best of three tests that were 95% compatible with each other was selected and recorded. Forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), Tiffeneau ratio (FEV1/FVC) and peak expiratory volume (PEF) (L/min) values were measured and both the measured values and the percentages of expected values were recorded.
Measurement of Respiratory Muscle Strength | 8 weeks
  Respiratory muscle strength was measured in accordance with ATS/ERS criteria using an electronic and portable intraoral pressure measuring device.All of the measurements were made in the sitting position with the feet in full contact with the ground. Nasal breathing was blocked with a nose clip. In order to measure the maximum inspiratory pressure (MIP), maximum expiratory maneuver was performed before the patient took the mouthpiece of the device into his mouth, and then maximal inspiration (Müller maneuver) was performed at maximum speed for 1-3 seconds. For maximum expiratory pressure measurement, the maximum inspiratory maneuver was performed before the mouthpiece of the device was taken into the mouth, and then maximal expiration (Valsalva maneuver) was performed at maximum speed for 1-3 seconds. 3 measurements were repeated for each evaluation and the highest value was recorded in "cmH2O".
Measurement of Functional Capacity | 8 weeks
  Functional capacity was measured with the 6-Minute Walk Test (6MWT) according to the guideline of ERS. The 6MWT to be a reliable, reproducible, and valid functional test for assessing exercise tolerance and endurance. Subjects were instructed to walk from one end to the other of a 30 m hallway at their own pace, while attempting to cover as much ground as possible in the allotted 6 min. The test was self-paced and the subject could rest if he or she so wished.
Measurement of Quality of Life | 8 weeks
  To determine the patients' quality of life, the Pediatric Quality of Life Scale (PedsQL 4.0), developed by Varni et al. and adapted into Turkish for the 8-12 age group by Sönmez and Başbakkal and its validity and reliability study was performed. The validity and reliability study of the 13-18 age group form of the scale was performed by Mermik et al. The total score that can be obtained from the 5-option Likert-type scale varies between 0 and 100, and scores closer to 0 indicate negative (bad) quality of life, while scores closer to 100 indicate positive (good) quality of life.
Measurement of Fatigue | 8 weeks
  The Brief Fatigue Inventory (BFI), developed by Mendoza et al. for cancer patients and whose Turkish validity and reliability study was conducted by Çinar et al., was used to determine the fatigue levels of the participants. The inventory evaluates the fatigue level of the patients in the last 24 hours and its effect on daily life activities (general activity, mood, walking ability, work life, relationships with other people, joy of life). The inventory consists of a total of 9 items, 3 of which measure general fatigue and 6 of which evaluate the effect of fatigue on daily life. The evaluation of the items is made by summing the scores between "0" (no fatigue at all) and "10" (the most severe fatigue you can experience), with "0" being the lowest score and "90" being the highest score. A low score indicates a low fatigue level and a high score indicates a high fatigue level. In this study, the evaluation was made based on the total score obtained from the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Semiramis Özyılmaz, Assoc. Prof., Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)